CLINICAL TRIAL: NCT00881959
Title: Multi-center, Post-market, Prospective, Randomized, Examiner-Only-Masked Study of Root Coverage With Acellular Dermal Matrix: Puros® Dermis Versus Alloderm®
Brief Title: Study of Root Coverage With Acellular Dermal Matrix: Puros® Dermis Versus Alloderm®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Zimmer Dental (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-800
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Gingival Recession
Keywords: exposed Root Surface or Tooth; Tooth Sensitivity Miller Class I; Miller Class II; Gingival Margin
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Puros Dermis (Experimental): Experimental treatment group of subjects who each have a single non-adjacent Miller's Class I or II gingival recession defect, greater than or equal to 2 mm, located on the buccal aspect of the maxillary incisor, canine, or premolar.
  Interventions: Device: Puros® Dermis versus Alloderm®
- Group 2: Alloderm (Active Comparator): Control group of subjects who each have a single non-adjacent Miller's Class I or II gingival recession defect, greater than or equal to 2 mm, located on the buccal aspect of the maxillary incisor, canine, or premolar.
  Interventions: Device: Puros® Dermis versus Alloderm®

INTERVENTIONS:
Device: Puros® Dermis versus Alloderm® — Puros Dermis and Alloderm (both Allograft Tissue Matrix)
  Other Names: Allograft Tissue Matrix, Human Acellular Dermal Matrix (ACDM)

SUMMARY:
The purpose of the study is to evaluate whether clinical parameters for Puros Dermis are, at minimum, equivalent when compared to AlloDerm, the current industry standard, for the treatment of single, non-adjacent Miller's Class I or II gingival recession.

DETAILED DESCRIPTION:
This is a prospective, Post-market, Randomized, Examiner-Only Masked multi-center study to evaluate whether clinical parameters for Puros Dermis are at minimum, equivalent when compared to Alloderm, the current industry standard for the treatment of single, non-adjacent Miller's Class I or II gingival recession.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any ethnicity, between 18 and 99 years of age.
* No known allergies to study material.
* Able to communicate with the investigator and read, understand, and sign the informed consent form.
* Maxillary incisor, canine, or premolar with at least one Miller's Class I or II gingival recession defects that are not adjacent to one another.
* Depth of the gingival recession defects of 2mm or greater.
* No gingival surgery within the past 12 months at the defect site. No prior antibiotic use within 3 months with less than 2 weeks durations.
* Ability to maintain good oral hygiene.

Exclusion Criteria:

* Patients taking any medications known to cause gingival enlargement.
* Patients with unstable systemic diseases.
* Patients with compromised immune systems or unstable bleeding disorders.
* Patients with active infectious diseases (e.g. hepatitis, tuberculosis, HIV, etc.).
* Patients with a mental disability that may hinder participation in the study (e.g. inability to follow through with oral hygiene instructions, postoperative instructions, follow-up commitments, etc.).
* Patients taking steroid medications.
* Tobacco use or smoking within 1 year of screening visit (e.g. cigarettes, pipes, cigars, chew).
* Pregnant females or females attempting to get pregnant.
* Other conditions the investigator feels would inhibit from a good candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - University of Rochester, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 08 25 2009 to 04 24 2011. Subjects had a single non-adjacent Miller's class I or II gingival recession defect, greater than or equal to 2mm, located on the buccal aspect of the maxillary incisor, canine, or premolar. Subjects for this study were recruited from the PI's clinic.
Pre-assignment Details: Randomized
Groups:
- Arm 1: Puros Dermis: Subjects with a single non-adjacent Miller Class I or II gingival recession treated with Puros Dermis.
- Arm 2: Alloderm: Subjects with a single non-adjacent Miller Class I or II gingival recession treated with Alloderm.
Period: Overall Study
Arm/Group | Arm 1: Puros Dermis | Arm 2: Alloderm
Started | 38 | 42
Completed | 36 | 38
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Puros Dermis | Group 2: Alloderm | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 38 | 75
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.7) | 47.4 (14) | 46.4 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 10 | 16 | 26
Region of Enrollment [Number; unit: participants]
  United States | 38 | 42 | 80

OUTCOME MEASURES:

1. Primary Outcome: Non -Inferiority of Dermis to Alloderm
Description: Non -inferiority of Dermis to Alloderm will be assessed by comparison of the average change (from the preoperative value) in gingival recession measured at 12 months between defects receiving Puros Dermis and those receiving Alloderm.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm 1: Puros Dermis | Arm 2: Alloderm
Number analyzed (Participants) | 38 | 36
mm | 2.06 (1.11) | 2.00 (0.87)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm 1: Puros Dermis | Arm 2: Alloderm
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 2/38 | 0/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Puros Dermis (N=38) | Arm 2: Alloderm (N=42)
Infection, Other (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less